CLINICAL TRIAL: NCT03314701
Title: Biphasic Intermittent Positive Airway Pressure (BIPAP) Versus Airway Pressure Release Ventilation (APRV) in Patients With Multiple Fracture Ribs
Brief Title: Mechanical Ventilation in Multiple Fracture Ribs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sayed Kaoud Abd-Elshafy, Associate Professor of Anesthesiology and Critical Care, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB0000879659
Record Dates: First submitted 2017-10-14; First posted 2017-10-19 (Actual); Last update posted 2018-07-09 (Actual); Status verified 2018-07

CONDITIONS: Mechanical Ventilation
Keywords: Resting Energy Expenditure; Multiple Fracture Ribs; Ventilation
MeSH Terms: conditions — Respiratory Aspiration | interventions — Intermittent Positive-Pressure Ventilation; Continuous Positive Airway Pressure

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Active Comparator): Biphasic Intermittent Positive Airway Pressure (BIPAP) group:
  Following endotracheal intubation BIPAP mode will be started with:
  * Inspiratory positive airway pressure [IPAP] at 20 cmH2O
  * Expiratory positive airway pressure [EPAP] at 5 cmH2O
  * PRESSURE SUPPORT is difference between these two pressures [IPAP]- [EPAP]
  * Mandatory pressure will be delivered at rate of 10-12/min. To produce an end tidal carbon dioxide partial pressure in the range of 35-40 mmHg hypercapnia will not be allowed
  Interventions: Device: Biphasic Intermittent Positive Airway Pressure (BIPAP)
- Group 2 (Active Comparator): Airway Pressure Release Ventilation (APRV) group:
  * high airway pressure (Phigh) will be set at 20 cmH2O
  * low airway pressure ( Plow) will be set at 5 cmH2O
  * the release phase setting will be adjusted to terminate the peak expiratory flow rate to ≥ 50%; release frequency of 10-12 cycles/min
  * T high at 4.5-6 seconds
  * T low at 0.5 to 0.8 second
  Interventions: Device: Airway Pressure Release Ventilation (APRV)

INTERVENTIONS:
Device: Biphasic Intermittent Positive Airway Pressure (BIPAP) — Following endotracheal intubation BIPAP mode will be started with:
  * Inspiratory positive airway pressure [IPAP] at 20 cmH2O
  * Expiratory positive airway pressure [EPAP] at 5 cmH2O
  * PRESSURE SUPPORT is difference between these two pressures [IPAP]- [EPAP]
  * Mandatory pressure will be delivered at rate of 10-12/min. To produce an end tidal carbon dioxide partial pressure in the range of 35-40 mmHg hypercapnia will not be allowed
  Arms: Group 1
Device: Airway Pressure Release Ventilation (APRV) — * high airway pressure (Phigh) will be set at 20 cmH2O
  * low airway pressure ( Plow) will be set at 5 cmH2O
  * the release phase setting will be adjusted to terminate the peak expiratory flow rate to ≥ 50%; release frequency of 10-12 cycles/min
  * T high at 4.5-6 seconds
  * T low at 0.5 to 0.8 second
  Arms: Group 2

SUMMARY:
Chest trauma is the most common injury in the emergency trauma and rib fractures is the most common trauma in chest trauma. Severe rib fractures can cause paradoxical respiration and mediastinal swing, which has large effects on respiratory and circulatory system, result in acute respiratory distress syndrome. Mechanical ventilation can significantly improve the hypoxemia of the patients, correct paradoxical respiration, and treat the pulmonary atelectasis

DETAILED DESCRIPTION:
To compare between Biphasic Intermittent Positive Airway Pressure (BIPAP) ventilation and Airway Pressure Release Ventilation (APRV) mode in patients with multiple fracture ribs as regard:

* Resting Energy Expenditure
* Oxygenation
* Stability of Physiological Status as cardiovascular activity
* cardiac output
* arterial blood gas measurement including [ blood PH, arterial oxygen tension, arterial carbon dioxide tension, bicarbonate level and base deficit]
* lung and chest compliance
* Length of intensive care unit stay.
* The ICU mortality rate.
* The development of major complications as nosocomial infection (hospital acquired pneumonia and ventilator associated pneumonia), major atelectasis and pneumothorax.

ELIGIBILITY:
Inclusion Criteria:

• Isolated chest trauma patient with Multiple fracture ribs patients [ >3 ribs] who will be admitted to the surgical ICU for ventilatory support and will be expected to continue for 2 days or longer

Exclusion Criteria:

* Age < 18 years old.
* Pregnant patient.
* Patient who will require fraction of inspired oxygen more than 0.6.
* Air leak from the chest tube.
* Patient with body temperature > 39 Celsius.
* Acute hepatitis or severe liver disease (Child-Pugh class C).
* Left ventricular ejection fraction less than 30%.
* Heart rate less than 50 beats/min.
* Second or third-degree heart block.
* Systolic pressure < 90 mmHg despite of infusion of 2 vasopressors.
* Patients with known endocrine dysfunction.
* Patient with hypothermia
* Patient on Positive end expiratory pressure more than 14 cmH2o

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-10-25 (Actual); Primary Completion 2018-10 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Duration of mechanical ventilation | within one month
  The total duration of ventilatory support in both groups from randomization to successful weaning (hours)

SECONDARY OUTCOMES:
Resting Energy Expenditure | within the first 48 hours
  Energy expenditure will be measured using indirect calorimetry via a metabolic module on General Electric ventilator [CARESCAPE R860]
Physiological dead space | within the first 48 hours
  Physiological dead space will be measured in the two groups after 30 minutes by Volumetric capnography which is included in the metabolic module on General Electric ventilator

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Asyut, Egypt